CLINICAL TRIAL: NCT05765344
Title: A Phase 1, Open-label, Parallel-group, Multiple-dose Study to Evaluate the Pharmacokinetics of Bulevirtide in Participants With Normal and Impaired Hepatic Function
Brief Title: Study of Bulevirtide in Participants Who Have Normal or Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-589-6162
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Impairment; Healthy
MeSH Terms: interventions — bulevirtide; myrcludex-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group A: Bulevirtide (BLV) 2 mg, Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment will receive BLV 2 mg subcutaneous (SC) injection, once daily for 6 days starting on Day 1.
  Interventions: Drug: Bulevirtide
- Group A: BLV 2 mg, Matched Control (Experimental): Control group participants with normal hepatic function matched similar to moderate hepatic impairment participants will receive BLV 2 mg SC injection once daily for 6 days starting on Day 1.
  Interventions: Drug: Bulevirtide
- Group B: BLV 2 mg, Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment will receive BLV 2 mg SC injection, once daily for 6 days starting on Day 1.
  Interventions: Drug: Bulevirtide
- Group B: BLV 2 mg, Matched Control (Experimental): Control group participants with normal hepatic function matched similar to moderate hepatic impairment participants will receive BLV 2 mg SC injection once daily for 6 days starting on Day 1.
  Interventions: Drug: Bulevirtide
- Group C: BLV 10 mg, Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment will receive BLV 10 mg SC injection, once daily for 6 days starting on Day 1.
  Interventions: Drug: Bulevirtide
- Group C: BLV 10 mg, Matched Control (Experimental): Control group participants with normal hepatic function matched similar to moderate hepatic impairment participants will receive BLV 10 mg SC injection once daily for 6 days starting on Day 1.
  Interventions: Drug: Bulevirtide
- Group D: BLV 10 mg, Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment will receive BLV 10 mg SC injection, once daily for 6 days starting on Day 1.
  Interventions: Drug: Bulevirtide
- Group D: BLV 10 mg, Matched Control (Experimental): Control group participants with normal hepatic function matched similar to moderate hepatic impairment participants will receive BLV 10 mg SC injection once daily for 6 days starting on Day 1.
  Interventions: Drug: Bulevirtide

INTERVENTIONS:
Drug: Bulevirtide — 2 mg administered via subcutaneous injections.
  Other Names: Hepcludex®; Myrcludex B
  Arms: Group A: BLV 2 mg, Matched Control; Group A: Bulevirtide (BLV) 2 mg, Moderate Hepatic Impairment; Group B: BLV 2 mg, Matched Control; Group B: BLV 2 mg, Severe Hepatic Impairment
Drug: Bulevirtide — 10 mg administered via subcutaneous injections.
  Other Names: Hepcludex®; Myrcludex B
  Arms: Group C: BLV 10 mg, Matched Control; Group C: BLV 10 mg, Moderate Hepatic Impairment; Group D: BLV 10 mg, Matched Control; Group D: BLV 10 mg, Severe Hepatic Impairment

SUMMARY:
The goals of this study are to measure the amount of bulevirtide (BLV) that gets into the blood stream and how long it takes to get rid of it, measure the effect of BLV on bile acids, and evaluate the safety and tolerability of multiple doses of BLV in participants with normal and impaired hepatic (liver) function.

ELIGIBILITY:
Key Inclusion Criteria:

All individuals:

* Body mass index (BMI) of 18 ≤ BMI ≤ 40 kg/m^2 at screening.
* Have a calculated creatinine clearance (CLcr) of at least 60 mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at screening.
* Individuals assigned male at birth and individuals assigned female at birth and of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception as described in the protocol.
* Individuals have not donated blood within 56 days of study entry or plasma within 7 days of study entry and must refrain from blood donation from clinic admission, throughout the study period, and continuing for at least 30 days following the last dose of study drug.
* 12-lead electrocardiogram (ECG) evaluations at screening must be without clinically significant abnormalities as assessed by the investigator.
* Aside from hepatic impairment among the individuals with hepatic impairment, the individual must, in the opinion of the investigator, be sufficiently healthy for study participation based upon medical history, physical examination, vital signs, and screening laboratory evaluations.
* Must be willing and able to comply with all study requirements.

Individuals With Hepatic Impairment:

* Have a diagnosis of chronic (> 6 months), stable hepatic impairment (moderate or severe based upon the Child-Pugh-Turcotte (CPT) classification system for moderate or severe hepatic impairment [CPT Class B or C, respectively]) with no clinically significant change in hepatic status (as determined by the investigator) within the 2 months (60 days) prior to screening.

  * Individuals with moderate or severe hepatic impairment must have a score of 7 to 9 or 10 to 15 on the CPT classification system at screening. If an individual's score changes during the study, the score at screening will be used for classification.
* Must meet all of the following laboratory parameters at screening:

  * alanine aminotransferase (ALT) ≤ 10 × upper limit of normal (ULN)
  * aspartate aminotransferase (AST) ≤ 10 × ULN
  * platelets ≥ 25,000/mm^3
  * hemoglobin ≥ 9 g/dL
* Individuals with hepatic impairment who have not been on a stable dose of concomitant medications for at least 4 weeks prior to screening (or 5 half-lives, whichever is longer) and/or for whom dose changes are likely to occur during the study should have their medications reviewed and approved by the sponsor.

Matched Control Individuals With Normal Hepatic Function:

* Have alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, international normalized ratio, and total bilirubin at or below the ULN; and albumin above the lower limit of normal at screening and at admission.
* Must be matched for age (± 10 years), sex (assigned at birth), and BMI (± 20%, 18 ≤ BMI ≤ 40 kg/m^2) with an individual in the hepatic impairment group.

Key Exclusion Criteria:

All Individuals:

* Positive serum pregnancy test at screening and at admission.
* Breastfeeding individual.
* Have received any study drug within 30 days prior to study dosing.
* Have current alcohol or substance abuse judged by the investigator to potentially interfere with individual compliance or individual safety, or a positive drug or alcohol test at screening or admission.
* Have poor venous access that limits phlebotomy.
* Have been treated with systemic steroids, immunosuppressant therapies, or chemotherapeutic agents within 3 months prior to screening or is expected to receive these agents during the study.
* Have a history of any of the following:

  * Significant serious skin disease, such as but not limited to rash, food allergy, eczema, psoriasis, or urticaria.
  * Significant drug sensitivity or drug allergy (such as anaphylaxis or hepatoxicity).
  * Known hypersensitivity to the study drugs, their metabolites, or to formulation excipients.
  * Significant cardiac disease (including history of myocardial infarction based on ECG and/or clinical history, any history of ventricular tachycardia, congestive heart failure, or dilated cardiomyopathy with left ventricular ejection fraction ≤ 40%); or a family history of long QT syndrome, or unexplained death in an otherwise healthy individual between the ages of 1 and 30 years.
  * Syncope, palpitations, or unexplained dizziness.
  * Implanted defibrillator or pacemaker.
* Have any serious or active medical or psychiatric illness (including depression).
* Requirement for ongoing therapy with or prior use of any prohibited medications listed in the protocol.

Individuals With Hepatic Impairment:

* Have a positive test result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody with detectable HCV ribonucleic acid (RNA) at screening.
* Suspicion of hepatocellular carcinoma (ie, if alpha-fetoprotein > 20 ng/mL at screening).
* Anticipated changes in concomitant medications or dosage used to treat symptoms of hepatic impairment or associated comorbid conditions that could lead to clinically significant changes in medical conditions during the study.
* Use of known hepatotoxic medications, clinical organic anion transporting polypeptide (OATP)1B1/3 inhibitors, or sodium-taurocholate cotransporting polypeptide (NTCP) inhibitors (half-maximal inhibitory concentration (IC50) or kinetic inhibition constant [Ki] < 20 μM).
* Positive test for drugs of abuse, including alcohol at screening or admission, with the exception of opioids and tetrahydrocannabinol (marijuana) under prescription and verified by the investigator as for pain management.

Matched Control Individuals With Normal Hepatic Function:

* Have a positive test result for HIV antibody, HBsAg, or HCV antibody.
* Have a history of liver disease including Gilbert's disease.
* Have taken any prescription medications or over-the-counter medications, including herbal products, within 28 days prior to start of study drug dosing, with the exception of vitamins and/or acetaminophen and/or ibuprofen and/or hormonal contraceptive medications.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (6):
  - Orange County Research Center, Lake Forest, California
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar P, Mercier RC, Nieves W, Pan D, Tseng S, Chee GM, et al. Pharmacokinetics, Pharmacodynamics, and Safety of Bulevirtide 2 mg Once Daily for 6 Days in Participants With Moderate and Severe HI and in Matched Control Participants With Normal Hepatic Function. American Association for the Study of Liver Diseases (AASLD); 1154: 15 November 2024
- [Background] Parag Kumar, Wildaliz Nieves, David Pan, Steve Tseng, Yuejiao Jiang, Yehong Wang, Ann Qin, Teckla Akinyi, Renee-Claude Mercier. Pharmacokinetics, Pharmacodynamics, and Safety of Bulevirtide 10 mg Once Daily for 6 Days in Participants With Moderate HI and in Matched Control Participants With Normal Hepatic Function. EASL - European Association for the Study of the Liver May 7-10, 2025 Amsterdam the Netherlands
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-589-6162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States.
Pre-assignment Details: 124 participants were screened.
Groups:
- Group A: Bulevirtide (BLV) 2 mg, Moderate Hepatic Impairment: Participants with moderate hepatic impairment received BLV 2 mg subcutaneous (SC) injection, once daily for 6 days starting on Day 1.
- Group A: BLV 2 mg, Matched Control; Group B: BLV 2 mg, Matched Control: Control group participants with normal hepatic function matched similar to moderate hepatic impairment participants received BLV 2 mg SC injection once daily for 6 days starting on Day 1.
- Group B: BLV 2 mg, Severe Hepatic Impairment: Participants with severe hepatic impairment received BLV 2 mg SC injection, once daily for 6 days starting on Day 1.
- Group C: BLV 10 mg, Moderate Hepatic Impairment: Participants with moderate hepatic impairment received BLV 10 mg SC injection, once daily for 6 days starting on Day 1.
- Group C: BLV 10 mg, Matched Control; Group D: BLV 10 mg, Matched Control: Control group participants with normal hepatic function matched similar to moderate hepatic impairment participants received BLV 10 mg SC injection once daily for 6 days starting on Day 1.
- Group D: BLV 10 mg, Severe Hepatic Impairment: Participants with severe hepatic impairment received BLV 10 mg SC injection, once daily for 6 days starting on Day 1.
Period: Overall Study
Arm/Group | Group A: Bulevirtide (BLV) 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Started | 11 | 11 | 8 | 8 | 10 | 10 | 8 | 8
Completed | 10 | 10 | 8 | 8 | 10 | 10 | 8 | 8
Not Completed | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug BLV.
Groups:
- Group A: BLV 2 mg, Moderate Hepatic Impairment: Participants with moderate hepatic impairment received BLV 2 mg SC injection, once daily for 6 days starting on Day 1.
- Total: Total of all reporting groups
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control | Total
Number analyzed (Participants) | 11 | 11 | 8 | 8 | 10 | 10 | 8 | 8 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 7 | 7 | 7 | 8 | 8 | 7 | 61
  >=65 years | 4 | 1 | 1 | 1 | 3 | 2 | 0 | 1 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (10.5) | 56 (7.4) | 47 (12.5) | 46 (12.7) | 61 (7.4) | 59 (6.0) | 52 (7.7) | 53 (8.6) | 55 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 4 | 3 | 3 | 3 | 3 | 26
  Male | 8 | 8 | 4 | 4 | 7 | 7 | 5 | 5 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 5 | 7 | 8 | 6 | 6 | 6 | 52
  Not Hispanic or Latino | 4 | 4 | 3 | 1 | 2 | 4 | 2 | 2 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 6
  White | 10 | 9 | 8 | 8 | 10 | 9 | 8 | 6 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 8 | 8 | 10 | 10 | 8 | 8 | 74

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of Bulevirtide (BLV)
Description: AUCtau was defined as the area under the concentration versus time curve (AUC) over the dosing interval at steady state.
Time Frame: Day 6: Predose and up to 24 hours postdose
Population: The plasma PK Analysis Set included all enrolled participants who took at least 1 dose of BLV and had at least 1 measurable plasma PK concentration data reported by PK laboratory for the analyte BLV. Participants in the plasma PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 9 | 7 | 8 | 5 | 10 | 10 | 8 | 8
h*ng/mL | 152 (110) | 150 (66.9) | 215 (71.7) | 113 (45.8) | 1270 (776) | 1560 (347) | 1520 (459) | 1600 (502)
Statistical Analysis 1: Comparison: Group A: BLV 2 mg, Moderate Hepatic Impairment vs Group A: BLV 2 mg, Matched Control; Test type: Other; Geometric least-squares mean ratio (%) = 87.2, 90% CI 2-sided [49.4 to 154] — ANOVA model with hepatic function as fixed effect was fitted to natural log-transformed values of the multiple dose PK parameter under evaluation. Geometric least-squares mean ratio (%) and 90%CI for hepatic impairment versus control were calculated
Statistical Analysis 2: Comparison: Group B: BLV 2 mg, Severe Hepatic Impairment vs Group B: BLV 2 mg, Matched Control; Test type: Other; Geometric least-squares mean ratio (%) = 197, 90% CI 2-sided [138 to 281] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group C: BLV 10 mg, Moderate Hepatic Impairment vs Group C: BLV 10 mg, Matched Control; Test type: Other; Geometric least-squares mean ratio (%) = 73.4, 90% CI 2-sided [54.4 to 99.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group D: BLV 10 mg, Severe Hepatic Impairment vs Group D: BLV 10 mg, Matched Control; Test type: Other; Geometric least-squares mean ratio (%) = 95.8, 90% CI 2-sided [73.1 to 126] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: PK Parameter: Cmax,ss of BLV
Description: Cmax,ss was defined as the maximum observed concentration of drug at steady state.
Time Frame: Day 6: Predose and up to 24 hours postdose
Population: Participants in the Plasma BLV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 10 | 8 | 8
ng/mL | 29.5 (23.8) | 22.7 (14.7) | 61.4 (27.6) | 15.2 (6.64) | 175 (113) | 261 (64.1) | 293 (96.8) | 263 (101)
Statistical Analysis 1: Comparison: Group A: BLV 2 mg, Moderate Hepatic Impairment vs Group A: BLV 2 mg, Matched Control; Test type: Other; Geometric least-squares mean ratio (%) = 117, 90% CI 2-sided [67.1 to 205] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group B: BLV 2 mg, Severe Hepatic Impairment vs Group B: BLV 2 mg, Matched Control; Test type: Other; Geometric least-squares mean ratio (%) = 401, 90% CI 2-sided [271 to 593] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group C: BLV 10 mg, Moderate Hepatic Impairment vs Group C: BLV 10 mg, Matched Control; Test type: Other; Geometric least-squares mean ratio (%) = 58.3, 90% CI 2-sided [40.8 to 83.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group D: BLV 10 mg, Severe Hepatic Impairment vs Group D: BLV 10 mg, Matched Control; Test type: Other; Geometric least-squares mean ratio (%) = 114, 90% CI 2-sided [80.7 to 161] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: PK Parameter: AUC0-24h of BLV
Description: AUC0-24h was defined as the partial area under the concentration versus time curve from time zero to time 24 hours.
Time Frame: Day 1: Predose and up to 24 hours postdose
Population: Participants in the Plasma BLV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 11 | 9 | 7 | 6 | 10 | 10 | 8 | 8
h*ng/mL | 82.9 (55.2) | 54.0 (12.8) | 174 (77.9) | 51.2 (8.90) | 672 (434) | 850 (337) | 1220 (350) | 750 (376)

4. Secondary Outcome: PK Parameter: Tmax of BLV
Description: Tmax was defined as the time (observed time point) of Cmax.
Time Frame: Days 1 and 6: Predose and up to 24 hours postdose
Population: Participants in the Plasma BLV PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 11 | 11 | 8 | 8 | 10 | 10 | 8 | 8
hours
  Day 1 | 1.50 [0.500 to 3.00] | 1.48 [1.00 to 2.00] | 1.00 [0.983 to 1.50] | 1.50 [1.00 to 2.03] | 4.00 [1.00 to 9.00] | 5.00 [2.00 to 9.00] | 3.00 [1.50 to 4.00] | 5.00 [1.50 to 9.00]
  Day 6: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 10 | 8 | 8
  Day 6 | 1.38 [0.500 to 1.60] | 1.51 [1.03 to 3.00] | 1.02 [1.00 to 1.50] | 1.75 [1.00 to 3.00] | 3.00 [3.00 to 6.00] | 3.00 [2.00 to 4.00] | 2.50 [2.00 to 3.00] | 3.00 [2.97 to 4.00]

5. Secondary Outcome: PK Parameter: Cmax of BLV
Description: Cmax was defined as the maximum observed plasma concentration of drug.
Time Frame: Day 1: Predose and up to 24 hours postdose
Population: Participants in the Plasma BLV PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 11 | 11 | 8 | 8 | 10 | 10 | 8 | 8
ng/mL | 23.7 (15.2) | 12.6 (4.28) | 57.7 (24.2) | 12.4 (3.84) | 99.2 (94.3) | 127 (65.6) | 230 (85.4) | 103 (69.6)

6. Secondary Outcome: PK Parameter: t1/2 of BLV
Description: t1/2 was defined as estimate of the terminal elimination half-life of the drug in plasma, calculated by dividing the natural log of 2 by the terminal elimination rate constant (λz).
Time Frame: Day 6: Predose and up to 48 hours postdose
Population: Participants in the Plasma BLV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 10 | 7 | 8 | 8 | 10 | 10 | 8 | 8
hours | 3.34 (1.31) | 2.86 (0.686) | 2.31 (0.791) | 5.05 (2.39) | 3.49 (1.15) | 2.80 (0.795) | 2.78 (0.750) | 3.33 (0.975)

7. Secondary Outcome: PK Parameter: CLss/F of BLV
Description: CLss/F was defined as the apparent clearance at the steady state (CLss) after administration of the drug:
  CLss/F = Dose/AUCtau, where "Dose" is the dose of the drug per interval.
Time Frame: Day 6: Predose and up to 48 hours postdose
Population: Participants in the Plasma BLV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 10 | 7 | 8 | 8 | 10 | 10 | 8 | 8
L/h | 22.1 (13.9) | 15.8 (7.21) | 9.97 (2.46) | 19.8 (7.20) | 9.63 (3.88) | 6.70 (1.62) | 7.06 (1.98) | 6.76 (2.10)

8. Secondary Outcome: PK Parameter: Vss/F of BLV
Description: Vss/F was defined as the apparent steady-state volume of distribution of the drug.
Time Frame: Day 6: Predose and up to 48 hours postdose
Population: Participants in the Plasma BLV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 10 | 7 | 8 | 8 | 10 | 10 | 8 | 8
liters | 119 (100) | 70.7 (46.3) | 34.4 (16.1) | 148 (78.8) | 52.6 (33.5) | 27.8 (13.9) | 28.4 (11.9) | 34.5 (19.4)

9. Secondary Outcome: Pharmacodynamic (PD) Parameter: Ctrough of Total Bile Acids (BA)
Description: Ctrough was defined as the concentration of total BA at the end of the dosing interval.
Time Frame: Predose on Days 2, 3, 4, 5, 7, and 8
Population: The plasma pharmacodynamic (PD) Analysis Set included all enrolled participants who received at least 1 dose of study drug BLV and had at least 1 measurable plasma PD concentration value reported for the analyte BA. Participants in the Plasma BA PD Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 10 | 8 | 8
uM
  Day 2 | 26.5 (27.1) | 4.68 (3.06) | 223 (131) | 5.18 (4.79) | 50.6 (55.1) | 25.7 (19.6) | 158 (60.5) | 31.0 (25.5)
  Day 3: number analyzed (Participants) | 10 | 10 | 7 | 8 | 10 | 10 | 8 | 8
  Day 3 | 46.3 (49.7) | 7.96 (7.00) | 213 (132) | 6.60 (2.74) | 67.2 (70.9) | 22.6 (9.53) | 180 (69.4) | 29.5 (25.1)
  Day 4 | 41.9 (50.5) | 6.86 (3.58) | 192 (121) | 6.03 (5.32) | 57.3 (46.0) | 23.3 (14.8) | 157 (87.1) | 16.1 (8.68)
  Day 5 | 30.5 (23.3) | 7.65 (3.85) | 201 (119) | 7.96 (6.01) | 50.6 (26.2) | 25.1 (12.2) | 176 (96.1) | 23.7 (13.9)
  Day 7 | 38.2 (37.3) | 10.2 (5.55) | 170 (91.3) | 8.44 (7.68) | 80.7 (65.9) | 21.8 (13.7) | 222 (97.0) | 25.9 (16.0)
  Day 8 | 33.4 (37.4) | 6.76 (5.62) | 151 (82.0) | 5.69 (3.73) | 37.1 (53.1) | 7.29 (3.73) | 129 (78.9) | 11.0 (9.21)

10. Secondary Outcome: PD Parameter: Cmax of Total BA
Description: Cmax was defined as the maximum observed concentration of total BA.
Time Frame: Days 1 and 6: Predose and up to 24 hours postdose
Population: Participants in the Plasma BA PD Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 9 | 10 | 8 | 8 | 10 | 10 | 8 | 8
uM
  Day 1 | 46.6 (61.4) | 15.6 (15.4) | 317 (156) | 13.1 (4.30) | 176 (99.7) | 145 (44.5) | 305 (40.9) | 150 (72.0)
  Day 6: number analyzed (Participants) | 9 | 9 | 8 | 8 | 10 | 10 | 8 | 8
  Day 6 | 124 (117) | 85.5 (42.2) | 318 (97.9) | 62.9 (44.6) | 343 (134) | 180 (35.8) | 370 (51.7) | 221 (78.9)

11. Secondary Outcome: PD Parameter: AUC0-24h of Total BA
Description: AUC0-24 was defined as the partial area under the concentration versus time curve from time "0" to time "24" hours for total BA.
Time Frame: Days 1 and 6: Predose and up to 24 hours postdose
Population: Participants in the Plasma BA PD Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: uM*h
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 9 | 10 | 8 | 8 | 10 | 10 | 8 | 8
uM*h
  Day 1 | 766 (1010) | 195 (174) | 5870 (2930) | 168 (69.5) | 2270 (1440) | 1690 (348) | 5130 (918) | 1760 (748)
  Day 6: number analyzed (Participants) | 9 | 9 | 8 | 8 | 10 | 10 | 8 | 8
  Day 6 | 1840 (1790) | 1000 (391) | 5680 (2010) | 720 (472) | 4640 (2010) | 2330 (527) | 6840 (1250) | 2920 (1150)

12. Secondary Outcome: PD Parameter: NetAUC of Total BA
Description: NetAUC was defined as the positive portion of area under the baseline-adjusted biomarker concentration versus time curve over the dosing interval.
Time Frame: Days 1 and 6: Predose and up to 24 hours postdose
Population: Participants in the Plasma BA PD Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: uM*h
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 9 | 10 | 8 | 8 | 10 | 10 | 8 | 8
uM*h
  Day 1 | 259 (345) | 133 (154) | 1790 (1430) | 113 (66.9) | 1880 (1020) | 1630 (334) | 2380 (781) | 1690 (731)
  Day 6: number analyzed (Participants) | 9 | 9 | 8 | 8 | 10 | 10 | 8 | 8
  Day 6 | 768 (773) | 925 (392) | 1880 (1120) | 657 (467) | 4210 (1410) | 2270 (542) | 4030 (1220) | 2850 (1140)

13. Secondary Outcome: PD Parameter: Tmax of Total BA
Description: Tmax was defined as the time (observed time point) of Cmax of total BA.
Time Frame: Days 1 and 6: Predose and up to 24 hours postdose
Population: Participants in the Plasma BA PD Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 9 | 10 | 8 | 8 | 10 | 10 | 8 | 8
hours
  Day 1 | 9.08 [-0.500 to 12.0] | 9.00 [6.00 to 23.5] | 7.50 [4.00 to 12.0] | 12.0 [6.00 to 24.7] | 12.0 [6.00 to 12.0] | 10.5 [6.00 to 12.1] | 12.0 [6.00 to 12.0] | 10.6 [9.00 to 12.0]
  Day 6: number analyzed (Participants) | 9 | 9 | 8 | 8 | 10 | 10 | 8 | 8
  Day 6 | 6.02 [1.50 to 12.0] | 9.00 [6.00 to 12.0] | 7.50 [6.00 to 12.0] | 10.5 [4.00 to 12.1] | 12.0 [6.00 to 12.0] | 9.00 [3.00 to 12.0] | 12.0 [6.00 to 12.1] | 10.5 [6.00 to 12.0]

14. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug and/or any AEs leading to premature discontinuation of study drug. If the AE onset date is the same as the date of study drug start date then the AE onset time must be on or after the study drug start time. If the AE onset time is missing when the start dates were the same, the AE were considered treatment emergent. An AE was any untoward medical occurrence in a clinical study participant administered a study drug that did not necessarily had a causal relationship with the treatment.
Time Frame: First dose date up to Day 6 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 11 | 11 | 8 | 8 | 10 | 10 | 8 | 8
percentage of participants | 27.3 | 9.1 | 25.0 | 12.5 | 20.0 | 20.0 | 25.0 | 25.0

15. Secondary Outcome: Percentage of Participants With Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment emergent. Grading categories are determined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 1: mild, Grade 2: moderate, Grade 3: severe or medically significant, Grade 4: life-threatening; Grade 5: Death.
Time Frame: First dose date up to Day 6 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
Number analyzed (Participants) | 11 | 11 | 8 | 8 | 10 | 10 | 8 | 8
percentage of participants
  Any Grade 1 or Higher | 63.6 | 63.6 | 100.0 | 62.5 | 90.0 | 90.0 | 75.0 | 50.0
  Grade 3 or 4 | 0.0 | 0.0 | 0.0 | 0.0 | 10.0 | 0.0 | 25.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to Day 6 plus 30 days
Description: All-cause Mortality: The All Enrolled Analysis Set included all participants who received a study participant identification number in the study after screening.
  Adverse Events: The Safety Analysis Set included all participants who took at least 1 dose of study drug BLV.
Arm/Group | Group A: BLV 2 mg, Moderate Hepatic Impairment | Group A: BLV 2 mg, Matched Control | Group B: BLV 2 mg, Severe Hepatic Impairment | Group B: BLV 2 mg, Matched Control | Group C: BLV 10 mg, Moderate Hepatic Impairment | Group C: BLV 10 mg, Matched Control | Group D: BLV 10 mg, Severe Hepatic Impairment | Group D: BLV 10 mg, Matched Control
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/8 | 0/8 | 0/10 | 0/10 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/8 | 0/8 | 0/10 | 0/10 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/11 | 1/11 | 2/8 | 1/8 | 2/10 | 2/10 | 2/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: BLV 2 mg, Moderate Hepatic Impairment (N=11) | Group A: BLV 2 mg, Matched Control (N=11) | Group B: BLV 2 mg, Severe Hepatic Impairment (N=8) | Group B: BLV 2 mg, Matched Control (N=8) | Group C: BLV 10 mg, Moderate Hepatic Impairment (N=10) | Group C: BLV 10 mg, Matched Control (N=10) | Group D: BLV 10 mg, Severe Hepatic Impairment (N=8) | Group D: BLV 10 mg, Matched Control (N=8)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT05765344/Prot_000.pdf
  • Statistical Analysis Plan (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT05765344/SAP_001.pdf